CLINICAL TRIAL: NCT05640570
Title: The Preventive Effectiveness of the Individualized Jade Wind-Barrier Herbal Tea Bag on the Common Cold in Elderly With Qi-deficiency Constitution (CCJWBT): A Pragmatic Randomized Controlled Trial
Acronym: CCJWBT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Chair Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HKBU JC 005
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Preventive Effectiveness; Elderly With Qi-deficiency Constitution; The Individualized Jade Wind-Barrier Herbal Tea Bag; Common Cold; Pragmatic Randomized Controlled Trial
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The individualized Jade Wind-Barrier Herbal Tea Bag (JWBT) arm (Experimental)
  Interventions: Drug: The individualized Jade Wind-Barrier Herbal Tea Bag
- Control arm (No Intervention)

INTERVENTIONS:
Drug: The individualized Jade Wind-Barrier Herbal Tea Bag — The individualized Jade Wind Barrier Herbal Tea Bag is composed of Astragali Radix (Zhi Huangqi) 4g, Saposhnikoviae Radix (Fangfeng) 2g, Atractylodes macrocephala Koidz (Baizhu) 2g, Nelumbinis Folium (Heye) 1g, Chrysanthemum morifolium Ramat (Juhua) 1g.
  Arms: The individualized Jade Wind-Barrier Herbal Tea Bag (JWBT) arm

SUMMARY:
Objectives

Based on the individualized Jade Wind-Barrier Herbal Tea Bag intake after randomization, to evaluate the relationship of the individualized Jade Wind-Barrier Herbal Tea Bag intake and the improvement of Qi-deficiency Constitution on the common cold-associated outcomes.

Specific Aims 1:

To compare the incidence and recurrence of the common cold by the individualized Jade Wind-Barrier Herbal Tea Bag intake strategies (intake 3-month individualized Jade Wind-Barrier Herbal Tea Bag vs. no intake throughout the same trial period) in the HK Qi-deficiency Constitution elderly.

Specific Aims 2:

To determine the immunological index(es) and function changes by the intake strategies (intake 3-month individualized Jade Wind-Barrier Herbal Tea Bag vs. no intake throughout the same trial period) on the common cold among HK Qi-deficiency Constitution elderly.

Specific Aims 3:

To assess the change in the reductive ratio of the total scores of the Clinical Features of the Qi-deficiency Constitution Questionnaire by the individualized Jade Wind-Barrier Herbal Tea Bag intake strategies (intake 3-month individualized Jade Wind-Barrier Herbal Tea Bag vs. no intake throughout the same trial period) in the HK Qi-deficiency Constitution elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 years old or above,
2. HK residents capable of consenting and have agreed to participate,
3. Meet the assessment criteria of Qi-deficiency Constitution in TCMECQ-C at screening,
4. The number of the incidence of the common cold ≥ 1 times/year,
5. Able to intake the individualized Jade Wind-Barrier Herbal Tea Bag and complete the trial-related records/questionnaires and also withdraw blood.

Exclusion Criteria:

1. Not fulfilling the above inclusion criteria,
2. Not assessed to be Qi-deficiency Constitution,
3. Having serious mental and behavioral disorders that are unable to intake the individualized Jade Wind-Barrier Herbal Tea Bag, complete the trial-related records/questionnaires and withdraw blood,
4. Having neurological disorders such as dementia etc. that are unable to intake the individualized Jade Wind-Barrier Herbal Tea Bag and complete the trial-related records/questionnaires and withdraw blood,
5. Having serious diseases with undesirable conditions that are unable to intake the individualized Jade Wind-Barrier Herbal Tea Bag and complete the trial-related records/questionnaires and withdraw blood,
6. Other conditions that are unable to intake the individualized Jade Wind-Barrier Herbal Tea Bag and complete the trial-related records/questionnaires and withdraw blood,
7. Allergic to Chinese Herbal Medicine (Astragali Radix (Zhi Huangqi), Saposhnikoviae Radix (Fangfeng), Atractylodes macrocephala Koidz (Baizhu), Nelumbinis Folium (Heye), Chrysanthemum morifolium Ramat (Juhua)),
8. Taking Chinese Herbal Medicine or drugs to manage their health problems within two weeks and cannot stop the treatment during the study,
9. Have an abnormal liver and renal function analyzed results after randomization at screening.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 304 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Change in the incidence rate of the common cold from baseline (week 0) to the end of the intervention (week 13). | Around 30 minutes is needed to fill in both TCM Body Constitution Questionnaire (For Elderly People) (Cantonese version) (TCMECQ-C) and the Incidence of Common Cold Record (if participants catch cold).
  Comparing Q14 incidence frequency of the common cold in the TCM Body Constitution Questionnaire (For Elderly People) (Cantonese version) (TCMECQ-C) with Q4 incidence days (convert to incidence frequency) of the common cold in the Incidence of Common Cold Record (if participants catch cold).
Change in the reductive ratio of the total score of CFQCQ among the HK Qi- deficiency Constitution elderly from baseline (week 0) to the end of intervention (week 13). | Around 30 minutes is needed to fill in both the baseline and after intervention CFQCQ.
  Comparing the difference between the baseline score of the Clinical Features of the Qi-deficiency Constitution Questionnaire (CFQCQ) and the after intervention score of the CFQCQ.

SECONDARY OUTCOMES:
Changes in the persistence time of incident common cold among the HK Qi-deficiency Constitution elderly from baseline (week 0) to the end of intervention (week 13). | Around 30 minutes is needed to fill in both the baseline and after intervention Incidence of Common Cold Record (if participants catch cold).
  Comparing the difference between 1st month with the 3rd month on Q4 number of incidence days of the common cold (persistence time of incident common cold) in the Incidence of Common Cold Record (if participants catch cold).
Change in intervention index of the total score of TCMSSM among the HK Qi-deficiency Constitution elderly (if catch cold) from baseline (week 0) to the end of intervention (week 13). | Around 30 minutes is needed to fill in both the baseline and after intervention TCMSSM.
  Comparing the difference between the baseline and after intervention's intervention index of the total score of the Traditional Chinese Medicine Syndrome Scoring Method Questionnaire (TCMSSMQ).
Changes in the ranges of immune markers (Ig G, Ig A and Ig M) function analysis from baseline (week 0) to the end of intervention (week 13). | Around one month respectively to complete the baseline and after trial blood withdrawal. Another one month for the corresponding ELISA test on IgG, IgA and IgM.
  Comparing the difference between the ranges of immune markers (IgG, IgA and IgM) function analysis from baseline (week 0) to the end of intervention (week 13).

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-xiang Bian, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- School of Chinese Medicine, Hong Kong Baptist University, Hong Kong, Hong Kong, China